CLINICAL TRIAL: NCT05196594
Title: Analysis of the Intestinal Microbiome of Patients With Transthyretin Amyloidosis
Brief Title: Analysis of the Instestinal Microbiome of Patients With Transthyretin Amyloidosis
Acronym: AMIAT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 04456582
Record Dates: First submitted 2021-10-06; First posted 2022-01-19 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2021-10

CONDITIONS: Amyloidosis, Hereditary, Transthyretin-Related; Microbial Colonization
Keywords: gut microbiome
MeSH Terms: conditions — Amyloidosis, Hereditary, Transthyretin-Related; Communicable Diseases | interventions — Genetic Testing

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Feces
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Affected group by transthyretinal amyloidosis with cardiac involvement: collection of stools
  Interventions: Diagnostic Test: collection of stools for genetic analysis
- Affected group by transthyretinal amyloidosis without cardiac involvement: collection of stools
  Interventions: Diagnostic Test: collection of stools for genetic analysis
- healthy control group: collection of stools
  Interventions: Diagnostic Test: collection of stools for genetic analysis

INTERVENTIONS:
Diagnostic Test: collection of stools for genetic analysis — Intestinal microbiome analysis

SUMMARY:
Amyloidosis is a serious systemic disease. Cardiac involvement has a great impact on prognosis and can occur in its three main forms: acquired monoclonal light chain, hereditary transthyretinal and senile form. The physiopathogenesis basically results from the deposition of an abnormal protein (amyloid) with toxic properties to the myocyte. The scope of this study will be a hereditary transthyretinal amyloidosis (hATTR). It is known that amyloidotic cardiomyopathy due to transthyretin deposit is an underdiagnosed cause of heart failure in adults, being an important differential diagnosis of diseases that manifest with increased myocardial thickness, such as hypertrophic cardiomyopathy or myocardial hypertrophy that accompanies the different degrees of aortic valve stenosis.

The human gut microbiota is immensely diverse. It is estimated at around 100 trillion microorganisms, including bacteria, fungi and viruses. The microbiota of each individual is unique and determined by genetic factors such as age, type of delivery, use of antibiotics and diet. Recent data point to the hypothesis that the resilience of the intestinal microbiota plays a role in the process of disease development and health restoration.

DETAILED DESCRIPTION:
The scope of this study will be hereditary transthyretinal amyloidosis (hATTR). It is known that amyloidotic cardiomyopathy due to transthyretin deposition is an underdiagnosed cause of heart failure in adults, being an important differential diagnosis of diseases that manifest with increased myocardial thickness, such as hypertrophic cardiomyopathy or the myocardial hypertrophy that accompanies the different degrees of aortic valve stenosis.

The transthyretin protein is synthesized and secreted into the bloodstream mainly by the liver. Other organic sites also produce and secrete it in smaller amounts. The choroid plexus produces and releases transthyretin in the cerebrospinal fluid, while the cells of the pigmented retinal epithelium are also capable of producing and releasing it into the vitreous body. Formerly called prealbumin, transthyretin is composed of four monomers that circulate in tetrameric form. It has the main function of carrying retinol and thyroxine . The degeneration of the protein tetramer and its deposition in the different fluids in which it is present determine the clinical dysfunction and the specific phenotypes of ATTR.

The gene that decodes the transthyretin protein (TTR) is located on chromosome 18. In ATTRh, alterations in the amino acid sequence destabilize the tetramer. It is conventional to designate genetic variants by the initials of the normal amino acid followed by their position in the gene and the amino acid that replaces it. Thus, the Val30Met variant translates that methionine is in place of valine at position 30.

The cuminal event of the pathophysiology is the degeneration of the tetramer into monomers that, once denatured, infiltrate several structures in the form of amyloid fibrils. In the myocardium, this process causes rigidity and varying degrees of dysfunction secondary to the intrinsic toxicity of these fibrils and to the occupation of the interstitium.

Clinically, ATTR can manifest itself as an autonomic polyneuropathy or as a cardiomyopathy. Eventually, the phenotype can involve both manifestations . Changes in the cardiac conduction system and arrhythmias usually precede heart failure by years.

Within the spectrum of alterations resulting from autonomic neuropathy, different degrees of intestinal transit disorders may occur, manifested as diarrhea, constipation, nausea or even asymptomatically.

Digestive symptoms are one of the most relevant and early clinical aspects of amyloidotic polyneuropathy, due to their frequency and intensity and the negative influence they have on the well-being of patients. Important changes in gastrointestinal motility are the main justification for these manifestations, being an expression of neurovegetative dysautonomia. Occurs: diarrhea, constipation, nausea, vomiting and feeling of gastric fullness.

Weight loss is a progressive and important feature, usually early and constant. It may be linked to gastrointestinal manifestations, malabsorption or renal and digestive protein losses. It is one of the worst prognosis manifestations of the disease.

The human gut microbiota is immensely diverse. It is estimated at around 100 trillion microorganisms, including bacteria, fungi and viruses. The microbiota of each individual is unique and determined both by genetic factors and by age, type of delivery, use of antibiotics and diet. There is evidence that such microorganisms play a fundamental role in food digestion, vitamin synthesis, production of short-chain fatty acids, modulation of the immune system and protection against infections. In healthy individuals, bacteria of the phyla Firmicutes and Bacterioidetes usually predominate, followed by Verrucromicrobia and Actinobacteria. However, the relative proportions and species present can vary widely between individuals and fluctuate over time, particularly during the early stages of life and during the evolution of certain diseases. Recent data point to the hypothesis that the resilience of the intestinal microbiota plays a role in the process of disease development and health restoration.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of transthyretin amyloidosis documented by pathogenic transthyretin mutation;
* evidence of cardiac involvement on echocardiogram or MRI; amyloid deposit confirmed by Congo red staining or presence of myocardial scintigraphy with grade 2 or 3 uptake (with distant monoclonal gammopathy of uncertain significance (MGUS);
* in the presence of MGUS it is necessary to confirm the TTR protein in the tissue by immunohistochemistry or mass spectrometry. Non-consanguineous living with patients;
* Sign an informed consent form.

Exclusion Criteria:

* Inflammatory bowel disease or persistent diarrhea for more than two weeks;
* Use of antibiotics and/or prebiotic or probiotic supplements in the two months prior to collection;
* Concurrent participation in other clinical studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Three groups of patients: a group affected by transthyretinal amyloidosis with cardiac involvement, another group affected by transthyretinal amyloidosis but without cardiac involvement, and a third healthy control group who live and share eating habits similar to those of the patients.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Gut Microbiome | 12 months
  Gene number (diversity index)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Sao Paulo Medical School - The Heart Institute, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided